CLINICAL TRIAL: NCT02448693
Title: Randomised Tandem Colonoscopy of Narrow Band Imaging (NBI) and White Light Endoscopy in Patients With Endoscopic Piecemeal Mucosal Resection
Brief Title: Study of Narrow Band Imaging in the Characterization of Residual Neoplasia After Endoscopic Piecemeal Mucosal Resection
Acronym: CROMOPIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Fausto Riu, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CROMOPIE
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasms
Keywords: endoscopic mucosal resection; piecemeal polypectomy scar; colorectal neoplasms; Narrow Band Imaging; chromoendoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WLE-NBI (Experimental): Participants will be evaluated by same endoscopist, tandem colonoscopy. It consists of two revisions of the polypectomy scar using firstly High Definition White Light Endoscopy (WLE) and secondly Narrow Band Imaging. All suspected neoplasia will be classified macroscopically and resected and differentiated from both techniques. The rest of the gut will be inspected following conventional standards.
  Interventions: Device: WLE; Device: NBI
- NBI-WLE (Experimental): Participants will be evaluated by same endoscopist, tandem colonoscopy. It consists of two revisions of the polypectomy scar using firstly Narrow Band Imaging and secondly High Definition White Light Endoscopy (WLE). All suspected neoplasia will be classified macroscopically and resected and differentiated from both techniques. The rest of the gut will be inspected following conventional standards.
  Interventions: Device: WLE; Device: NBI

INTERVENTIONS:
Device: WLE — Evaluation of the polypectomy scar with High Definition White Light Endoscopy (WLE)
  Other Names: High Definition colonoscopy with White Light Endoscopy (WLE)
Device: NBI — Evaluation of the polypectomy scar with Narrow Band Imaging (NBI, Evis Exera III, Olympus).
  Other Names: Narrow Band Imaging

SUMMARY:
This study is designed to evaluate the diagnostic accuracy of Narrow Band Imaging (NBI) compared with High Definition White Light colonoscopy (WLE) for detection of residual neoplasia in subjects with piecemeal polypectomy scars.

DETAILED DESCRIPTION:
Resection of large sessile polyps in the colon (usually more than 2 cm) or those nonpolypoid neoplastic lesions (also called laterally spreading tumors or LST), confers technical difficulty and often are forced to remove into fragmented resection or endoscopic piecemeal mucosal resection. This has been associated with a recurrence of 25%. For this reason, clinical guidelines recommend endoscopic follow-up at 2 to 6 months after piecemeal resection of colorectal polyps to check for residual neoplasia.

Narrow-Band Imaging (NBI, Olympus) improves visibility and identification of the surface and vascular structures of colon polyps. In contrast to conventional chromoendoscopy, it is easily activated by pressing a button on the endoscope.

Virtual or conventional chromoendoscopy are applied during resection of polyps defining the border of the lesion. However, there are few studies using Narrow Band Imaging and do not allow to know whether the use of this technique could improve the detection of residual tumor after fragmented polypectomy and avoid complications, time and costs of biopsy and histological analysis.

In this context, the European Society of Gastrointestinal Endoscopy (ESGE) has recently published the first Guideline of Advanced Endoscopic Imaging for the Detection and Differentiation of Colorectal Neoplasia and recommends conventional or virtual chromoendoscopy in patients with piecemeal polypectomy scar (strong recommendation, low quality evidence).

The investigators will perform a randomised, controlled trial of tandem colonoscopy using NBI and WLE. The main goal is to compare the rate of detected neoplasia between both techniques and evaluate the diagnostic accuracy of NBI and WLE to histology as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who underwent a colonoscopy for any reason in the last 12 month
* Patients with a basal colonoscopy findings: ≥1 polyp removed in a piecemeal fashion regardless of the size

Exclusion Criteria:

* Diagnosis of a CRC in the basal colonoscopy
* Subjects who neglect to follow-up
* Subjects who do not accept informed consent
* Subjects with high risk of perforation or complications due to sedation, including patients with comorbidities (ASA IV-V)
* Inadequate bowel preparation for colonoscopy (defined by Boston Bowel Preparation Score (BBPS): ≤ 5 total points; or 0-1 points in any of the 3 segments of the colon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of residual neoplastic tissue detected with both techniques (NBI versus WLE) | less than 1 year after the basal colonoscopy
  Efficacy of NBI in detecting residual neoplasia compared with WLE

SECONDARY OUTCOMES:
Number of accurate detection of residual neoplastic tissue with morphologic features in both groups (NBI and WLE) compared with histopathology | less than 1 year after the basal colonoscopy
  Accuracy in detecting neoplastic tissue endoscopically compared with histopathology (gold standard)
Number of missed lesions on basal colonoscopy | less than 1 year after the basal colonoscopy
  Compare the number of missed lesions from the basal colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Riu, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooker JC, Saunders BP, Shah SG, Thapar CJ, Thomas HJ, Atkin WS, Cardwell CR, Williams CB. Total colonic dye-spray increases the detection of diminutive adenomas during routine colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2002 Sep;56(3):333-8. doi: 10.1016/s0016-5107(02)70034-5. PMID 12196768
- [Background] Kiesslich R, von Bergh M, Hahn M, Hermann G, Jung M. Chromoendoscopy with indigocarmine improves the detection of adenomatous and nonadenomatous lesions in the colon. Endoscopy. 2001 Dec;33(12):1001-6. doi: 10.1055/s-2001-18932. PMID 11740641
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] Khashab M, Eid E, Rusche M, Rex DK. Incidence and predictors of "late" recurrences after endoscopic piecemeal resection of large sessile adenomas. Gastrointest Endosc. 2009 Aug;70(2):344-9. doi: 10.1016/j.gie.2008.10.037. Epub 2009 Feb 27. PMID 19249767
- [Background] Atkin WS, Valori R, Kuipers EJ, Hoff G, Senore C, Segnan N, Jover R, Schmiegel W, Lambert R, Pox C; International Agency for Research on Cancer. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Colonoscopic surveillance following adenoma removal. Endoscopy. 2012 Sep;44 Suppl 3:SE151-63. doi: 10.1055/s-0032-1309821. Epub 2012 Sep 25. PMID 23012119
- [Background] Lieberman DA, Rex DK, Winawer SJ, Giardiello FM, Johnson DA, Levin TR. Guidelines for colonoscopy surveillance after screening and polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2012 Sep;143(3):844-857. doi: 10.1053/j.gastro.2012.06.001. Epub 2012 Jul 3. No abstract available. PMID 22763141
- [Background] Hurlstone DP, Sanders DS, Cross SS, Adam I, Shorthouse AJ, Brown S, Drew K, Lobo AJ. Colonoscopic resection of lateral spreading tumours: a prospective analysis of endoscopic mucosal resection. Gut. 2004 Sep;53(9):1334-9. doi: 10.1136/gut.2003.036913. PMID 15306595
- [Background] Rogart JN, Aslanian HR, Siddiqui UD. Narrow band imaging to detect residual or recurrent neoplastic tissue during surveillance endoscopy. Dig Dis Sci. 2011 Feb;56(2):472-8. doi: 10.1007/s10620-010-1289-z. Epub 2010 Jun 9. PMID 20532981